CLINICAL TRIAL: NCT01385631
Title: The Effect Of Ezetimibe In Addition To Optimal Cholesterol-Lowering Statin Therapy On The Plaque Composition In Patients With Acute Myocardial Infarction - Assessed By Optical Coherence Tomography And Intravascular Ultrasound.
Brief Title: Ezetimibe In Addition To Atorvastatin Therapy On The Plaque Composition In Patients With Acute Myocardial Infarction.
Acronym: OCTIVUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mikkel Hougaard, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OUH-OCTIVUS
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: ST-Segment Elevation Myocardial Infarction
Keywords: ST-Segment Elevation Myocardial Infarction; Intravascular ultrasound; IVUS; Optical coherence tomography; OCT; Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Randomized trial; Hypolipidemic Agents; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Enzyme Inhibitors; Lipid Regulating Agents; Therapeutic Uses
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin plus Placebo (Placebo Comparator): 50/100 patients are randomized to Atorvastatin 80 mg per day plus placebo.
  Interventions: Drug: Placebo
- Atorvastatin plus Ezetimibe (Experimental): 100 patients with ST elevation myocardial infarction are randomized 1:1 to either placebo or Ezetimibe 10 mg per day in addition to treatment with Atorvastatin 80 mg in both arms.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — 100 patients with ST elevation myocardial infarction are randomized 1:1 to either placebo or Ezetimibe 10 mg per day in addition to treatment with Atorvastatin 80 mg in both arms.
  Other Names: Ezetrol; Zarator
  Arms: Atorvastatin plus Ezetimibe
Drug: Placebo — 100 patients with ST elevation myocardial infarction are randomized 1:1 to either placebo or Ezetimibe 10 mg per day in addition to treatment with Atorvastatin 80 mg in both arms.
  Other Names: Ezetrol; Zarator
  Arms: Atorvastatin plus Placebo

SUMMARY:
The purpose of the study is to examine the effect of the cholesterol lowering agent Ezetimibe when used in addition to optimal treatment with Atorvastatin in patients with acute ST-Elevation Myocardial Infarction (STEMI) who have not been in prior statin therapy.

An area with arteriosclerosis not demanding intervention in a coronary vessel other than the infarct related is used as measuring point and is examined at time of the infarction and after 12 month using intravascular ultrasound and optical coherence tomography. At the same time the same techniques are used to examine the implanted stent.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) and intravascular ultrasound (IVUS) with tissue characterization (IVUS-TC) are relatively new expansions to intravascular assessments, and has the capacity to assess plaque composition and, potentially, to identify vulnerable plaques. One of the mechanisms by which statins improve patient outcomes may be by changing the composition of a "vulnerable" plaque. The main effect is believed to rely on a lowering of LDL-c. The question is whether a further reduction of LDL by adding ezetimibe to optimal cholesterol lowering therapy using statins may result in further plaque stabilization or reduction. This is the hypothesis of the current study.

100 patients are randomized to Ezetimibe 10 mg per day or placebo. All patients are treated with Atorvastatin 80 mg. OCT and IVUS are performed at inclusion (typically the day after Primary PCI) and again at follow-up after 12 month.

ELIGIBILITY:
Inclusion Criteria:

* ST segment elevation acute myocardial infarction
* 20% < angiographic diameter stenosis < 50% on a not previously revascularized native coronary artery
* Statin naïve
* In fertile women: Ongoing contraception with IUD or hormonal contraception.

Exclusion Criteria:

* Pharmacologic lipid lowering treatment before index hospitalization
* Atrial fibrillation, not well rate-controlled
* Ventricle frequency variation with more than a factor 2 over 1 minute
* Unconscious patients
* History of statin induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins) including Atorvastatin.
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception or have a positive serum pregnancy test (a serum-human chorionic gonadotrophin [Beta-HCG] analysis)
* History of malignancy (unless a documented disease free period exceeding 5-years is present) with the exception of basal cell or squamous cell carcinoma of the skin. Women with a history of cervical dysplasia would be permitted to enter the study provided they had 3 consecutive clear Papanicolaou (Pap) smears
* Uncontrolled hypothyroidism (TSH > 1.5xULN)
* Abnormal LFT's
* History of alcohol or drug abuse within the last 5 years (this may affect compliance)
* Current active liver disease (ALT/SGPT >2xULN or severe hepatic impairment (to protect patient safety as directed on the labels of currently approved statins)
* Unexplained creatine kinase (CK > 3xULN) (To protect patient safety) (will be increased at baseline because of acute ST segment elevation myocardial infarction a few days before enrolment)
* Serum creatinine >176mmol/L (2.0mg/dL) (unless the protocol specifically aims to investigate a chronic renal disease population)
* Participation in another investigational drug study less than 4 weeks before enrolment in the study, or according to subjects local ethics committee requirements where a larger period is stipulated (to avoid potential misinterpretation of overlapping adverse events)
* Treatments with cyclosporine
* Treatment with gemfibrozil

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Plaque volume and composition in a non-significant coronary plaque | After 12 months of follow-up
  Plaque volume assessed by intravascular ultrasound and Optical Coherence Tomography

SECONDARY OUTCOMES:
Change in plaque-composition (measured with Tissue Characterization) in a 10 mm segment of a native coronary vessel with a non-significant stenosis where plaque-volume at baseline is greatest. | After 12 months of follow-up
Change in percent of the plaque volume in the native coronary vessel with a non-significant stenosis. | After 12 months of follow-up
Change in percent of the plaque volume in the 10 mm segment of a native coronary vessel with a non-significant lesion where plaque volume at baseline is greatest. | After 12 months of follow-up
Change in absolute numbers of the plaque volume in the 10 mm segment of a native coronary vessel with a non-significant lesion where plaque volume at baseline is greatest. | After 12 months of follow-up
Change in percent of the plaque burden in the 10 mm segment of a native coronary vessel with a non-significant lesion where plaque volume at baseline is greatest. | After 12 months of follow-up
Change in percent of the plaque burden in a native coronary vessel with a non-significant lesion. | After 12 months of follow-up
Incomplete stent apposition. | After 12 months of follow-up
Edge response in stented segment. | After 12 months of follow-up
Stent expansion. | After 12 months of follow-up
Evaluation of the OCT-technique in clinical use compared to IVUS. | After 12 months of follow-up
Evaluation of the Resolute stents effect on neointima growth and apposition. | After 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Hougaard, MD, Principal Investigator — Department of Cardiology, Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense C, Denmark